CLINICAL TRIAL: NCT01739075
Title: Assessment of the Functional Significance of Coronary Stenoses Using Coronary CT-angiography and Non-invasive Fractional Flow Reserve Measurement.
Brief Title: Assessment of Coronary Stenoses Using Coronary CT-angiography and Non-invasive Fractional Flow Reserve Measurement.
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: M-5-12
Record Dates: First submitted 2012-11-27; First posted 2012-11-30 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2013-08

CONDITIONS: Myocardial Ischemia
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine whether a novel non-invasive method to estimate coronary blood flow (FFRct) is applicable to evaluate the functional significance of coronary stenoses in non-culprit vessels in a population of patients with recent STEMI (ST-elevation myocardial infarction) and multivessel disease. The diagnostic performance and reproducibility of FFRct as well as the qualitative and quantitative correlation between FFRct and the regional coronary blood flow will be examined.

DETAILED DESCRIPTION:
Coronary Computed Tomography Angiography (cCTA) is a non-invasive imaging modality that provides high-resolution images of coronary lesions. cCTA shows good diagnostic performance in detecting or excluding coronary artery stenoses, but the severity of the lesions is often overestimated. With invasive coronary angiography (ICA) the hemodynamic consequences of obstructive lesions can be estimated using Fractional Flow Reserve measurement (FFR). There is a good correlation between FFR and non-invasive ischemia tests such as stress echocardiography, exercise tolerance test or Single Photon Emission Computed Tomography (SPECT). Measurement of FFR during ICA represents the "gold standard" for assessment of the hemodynamic significance of coronary artery lesions. The major disadvantage of FFR is that it is an invasive measurement, and consequently there is a risk of complications. Recently a non-invasive method to determine FFR has been developed (FFRct). FFRct is performed using standard cCTA images, and is based on computational fluid dynamics. The hemodynamic consequence of stenotic lesions is determined at rest and under simulated condition of hyperemia.

Acute myocardial infarction (MI) is divided into STEMI and NSTEMI on the basis of ECG changes. In Denmark patients with STEMI are treated with primary percutaneous intervention (PPCI) of the culprit lesion. Any non-culprit lesions are typically assessed with FFR after 3-4 weeks.

Even though the rate of complications during ICA with FFR is low, these complications can be severe. Also the procedure is quite resource demanding. Thus it would be desirable if it in these patients could be non-invasively evaluated whether further revascularisation is indicated.

ELIGIBILITY:
Inclusion Criteria:

* Recent STEMI and indication for new ICA to assess non-culprit lesions

Exclusion Criteria:

* contraindications to adenosine
* allergy to contrast agent
* P-creatinine > 125 micromol/L
* atrial fibrillation
* age < 18 years
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with STEMI admitted at Aarhus Universtity Hospital and treated with primary PCI, and where the operater finds one or more residual stenoses in non-culprit vessels that needs to be assessed at a later time with ICA and FFR.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
FFRct measurement | Acute measurement
FFR measurement | Acute assessment

SECONDARY OUTCOMES:
Absolute regional myocardial perfusion | Acute assessment
  Assessed by cardiac Positron Emission Tomography (PET)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Gaur, MD, Principal Investigator — Aarhus University Hospital; Bjarne L Nørgaard, MD, Ph.D., Study Chair — Aarhus University Hospital
Locations (1):
- Department of Cardiology, Aarhus University Hospital, Skejby, Aarhus N, Denmark

REFERENCES:
- [Derived] Gaur S, Taylor CA, Jensen JM, Botker HE, Christiansen EH, Kaltoft AK, Holm NR, Leipsic J, Zarins CK, Achenbach S, Khem S, Wilk A, Bezerra HG, Lassen JF, Norgaard BL. FFR Derived From Coronary CT Angiography in Nonculprit Lesions of Patients With Recent STEMI. JACC Cardiovasc Imaging. 2017 Apr;10(4):424-433. doi: 10.1016/j.jcmg.2016.05.019. Epub 2016 Oct 12. PMID 27743953